CLINICAL TRIAL: NCT03506581
Title: Discovering Carbohydrate Metabolism Alterations in Normoglycemic Obese Patients Study
Brief Title: Dysfunctional Adiposity and Glucose Impairment
Acronym: DICAMANO
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: 167/2016
Record Dates: First submitted 2018-02-06; First posted 2018-04-24 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-02

CONDITIONS: Body Composition; Visceral Obesity; Carbohydrate Intolerance; Obesity, Abdominal; Cardiovascular Risk Factor; Beta-cell Function; Insulin Resistance; Oral Glucose Tolerance Test
MeSH Terms: conditions — Obesity, Abdominal; Glucose-Galactose Malabsorption; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a large and comprehensively phenotyped cohort with fasting glycaemia where the predictive value of body composition and anthropometric measures of total and central fat distribution for postprandial carbohydrate intolerance are studied.

DETAILED DESCRIPTION:
Subjects aged 18-70 years, who attended the Department of Endocrinology and Nutrition of the Clínica Universidad de Navarra from 2009-2014 for a check-up were offered to participate in the DICAMANO study. 853 subjects agreed to take part. Only those individuals with a normal fasting glucose level (≤5.5 mmol l-1) were analysed. Subjects with T2DM or severe renal, liver or thyroid dysfunction were excluded. Participants were instructed to temporarily discontinue for 48 hours any medication known to affect glucose or lipid metabolism. On the day of the study visit, each subject had a complete routine clinical assessment to evaluate the presence of cardiovascular, respiratory, renal or endocrine disorders. All patients underwent a 75-g OGTT with a concomitant anthropometric study, blood pressure monitoring and lipid profile analyses. They were classified by glucose tolerance on the basis of blood glucose levels according to ADA diagnostic criteria for T2DM (2017). Carbohydrate intolerance was defined as a 2-hOGTT glucose level ≥7.8 mmol l-1 (mg dl-1). Body composition, visceral adipose tissue, anthropometry study, OGTT-based parameters and cardiovascular risk factors are measured.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose level ≤ 5.5 mmol l-1
* BMI ≥ 25

Exclusion Criteria:

* Type 2 diabetes mellitus
* Severe renal, liver or thyroid dysfunction

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18-70 years, who attended the Department of Endocrinology and Nutrition of the Clínica Universidad de Navarra from 2009-2014 for a check-up were offered to participate in the DICAMANO study
Sampling Method: Probability Sample
Enrollment: 853 (Actual)
Dates: Start 2009-01-29 (Actual); Primary Completion 2014-08-28 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
Body fat percentage and carbohydrate intolerance | Baseline
  Investigate whether body fat percentage estimated by air-displacement plethysmography (Bod-Pod®, Life Measurements, Concord, CA, USA) predicts postprandial carbohydrate intolerance early on in the metabolic dysregulation process.
  Body fat percentage (BF%) is calculated from body density by means of the Siri equation.
Neck circumference as screening tool | Baseline
  Examine the predictive value of neck circumference as screening tool for the selection of patients who are most likely to benefit from an oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Waist-to-hip ratio as screening tool | Baseline
  Examine the predictive value of waist-to-hip ratio as screening tool for the selection of patients who are most likely to benefit from an oral glucose tolerance test (OGTT). Waist-to-hip ratio was calculated as waist circumference divided by hip circumference. Waist circumference was measured at the midpoint between the iliac crest and the rib cage on the mid-axillary line, and hip circumference at the level of the greater trochanters was measured to the nearest millimetre using a flexible tape.
Waist-to-height ratio as screening tool | Baseline
  Examine the predictive value of waist-to-height ratio as screening tool for the selection of patients who are most likely to benefit from an oral glucose tolerance test (OGTT). Waist-to-height ratio was calculated as waist circumference divided by height.
BMI as screening tool | Baseline
  Examine the predictive value of body adiposity index (BMI) as screening tool for the selection of patients who are most likely to benefit from an oral glucose tolerance test (OGTT). BMI was calculated as weight in kilograms divided by height in meters squared.
Body adiposity index as screening tool | Baseline
  Examine the predictive value of body adiposity index (BAI) ([hip circumference/height1.5]-18) as screening tool for the selection of patients who are most likely to benefit from an oral glucose tolerance test (OGTT).
Central fat depot and carbohydrate intolerance | Baseline
  Investigate whether central fat depot predicts postprandial carbohydrate intolerance early on in the metabolic dysregulation process. Visceral and abdominal adiposity was quantified by the use of the abdominal bioelectrical impedance analysis device ViScan (Tanita AB-140, Tanita Corp., Tokyo, Japan).
Central fat depot and cardiometabolic risk | Baseline
  Investigate whether a higher central fat depot is able to identify those individuals with higher inflammatory parameters (c-reactive protein, homocysteine and uric acid) and cardiovascular risk (higher rate of hypercholesterolemia, hypertension and/or obstructive sleep apnea).
  Body fat percentage (BF%) is calculated from body density by means of the Siri equation.
Body fat percentage and cardiometabolic risk | Baseline
  Investigate whether a higher body fat percentage is able to identify those individuals with higher inflammatory parameters (c-reactive protein, homocysteine and uric acid) and cardiovascular risk (higher rate of hypercholesterolemia, hypertension and/or obstructive sleep apnea).
  Body fat percentage (BF%) is calculated from body density by means of the Siri equation.
Prevalence of postprandial carbohydrate intolerance | Baseline
  Assess the prevalence of postprandial carbohydrate intolerance in individuals with normal fasting glycaemia
Oral glucose tolerance test parameters and cardiometabolic profile | Baseline
  Verification of the utility of the two-hour OGTT glucose value to select those individuals with higher cardiometabolic risk (higher rate of hypercholesterolemia, hypertension and/or obstructive sleep apnea).
Non-alcoholic fatty liver disease (NAFLD) and glucose dysregulation | Baseline
  Analyse the association between NAFLD and OGTT-based ß-cell function and insulin resistance in non-diabetic subjects.
OGTT-based indices as screening tool of NAFLD | Baseline
  Examine whether OGTT-based ß-cell function and insulin resistance indices could be used as screening tools for the selection of patients who are most likely to benefit from a NAFLD-study.
OGTT-derived glucose curve as screening tool of NAFLD | Baseline
  Examine whether the glucose response curve could be used as screening tool for the selection of patients who are most likely to benefit from a NAFLD-study.

CONTACTS AND LOCATIONS:
Overall Officials: Gema Frühbeck, PhD, Study Chair — Clínica Universidad de Navarra; Belén Pérez Pevida, MD, Principal Investigator — Clínica Universidad de Navarra

REFERENCES:
- [Derived] Perez-Pevida B, Nunez-Cordoba JM, Romero S, Miras AD, Ibanez P, Vila N, Margall MA, Silva C, Salvador J, Fruhbeck G, Escalada J. Discriminatory ability of anthropometric measurements of central fat distribution for prediction of post-prandial hyperglycaemia in patients with normal fasting glucose: the DICAMANO Study. J Transl Med. 2019 Feb 18;17(1):48. doi: 10.1186/s12967-019-1787-5. PMID 30777085